CLINICAL TRIAL: NCT04288583
Title: Bringing Parkinson Care Back Home
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-5845
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
Keywords: Wearable sensors; Falls; Physical activity; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SUMMARY

Rationale: For persons with Parkinson's disease (PD), medical decisions are based almost exclusively on periodic in-clinic evaluations by a neurologist or a nurse. For a variety of reasons, such "snapshots" are unable to capture the actual impact of PD on the patient's functioning in their own home environment. Outpatient evaluations cannot detect rare and typically domestic events, such as falls. In addition, episodic visits are not well suited to detect changes in important lifestyle issues, such as gradual declines in physical activity.

Objective: To objectively, continuously and accurately collect detailed information on (changes in) physical activity and fall patterns among patients with PD in daily life.

Study design: Observational cohort study in 200 patients with PD, with a 12 month follow-up period.

Study population: Patients with PD (n=200), with an increased fall risk (i.e. at least one fall within the last six months).

Intervention (if applicable): This study does not include an intervention. After a baseline assessment on demographics and PD symptoms, patients will use a remote monitoring system at home (a pendant falls detector) combined with an smartphone application aimed at falls self-reporting, and an application to report medication intake for 12 months. A similar set up (i.e.Vital@Home) has been previously tested on feasibility (Dossiernummer: 2017-3382). Additionally, patients will report sleep patterns through paper-based diaries.

Main study parameters/endpoints: The main study parameters are physical activity and number of falls. They are remotely registered by the pendant falls detector.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In this study, no invasive measurements will be performed. The participation is free of risks. Subjects could potentially benefit personally from participating in this study, as they can use the devices for free during the study and receive periodically feedback about physical activity and the occurrence of falls.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must confirm that they have been diagnosed with Parkinson's Disease by a neurologist (self-reported)
* Age 18 or older
* At least 1 fall incident in the previous 6 months. A fall is defined as any unexpected event that caused the person to unintentionally land on any lower surface (object, floor, or ground), regardless of any sustained injury (self-reported)
* Able and willing to provide written informed consent in accordance with Good Clinical Practice, and national and local regulation
* Fluent in Dutch

Exclusion Criteria:

* The patients receives advanced therapy for their Parkinson's disease (deep brain stimulation, duodopa pump, apomorphine pump);
* The patients shows cognitive of psychiatric impairments that may hinder successful completion of the study protocol (as judged by the researcher running the recruitment).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients diagnosed with Parkinson's disease with an increased fall risk (i.e. who reported at least one fall in the last 6 months).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Falls | Continuously over 12 months
  Number of alls measured with wearable sensors
Physical activity | Continuously over 12 months
  Minutes of physical activity performed during daily-life measured with wearable sensors

SECONDARY OUTCOMES:
Physical activity | Twice - baseline and after 12 months
  LASA physical activity questionnaire, in which the higher the score the better
Walking capacity | Once - baseline
  6-meter walking test, in which the higher the distance walked the better
Falls | Twice - baseline and after 12 months
  Falls history questionnaire
Functional lower extremity strength | Once - baseline
  Five-times-sit-to-stand, in which the faster the task is completed the better
Fear of falling | Twice - baseline and after 12 months
  Falls Efficacy Scale International, with scores ranging from 16 to 64 points, in which the a higher score indicates worse fear of falling
Compliance | Continuously over 12 months
  Number of days in which participants worn the device for more than 8 hours
Patients demographics | Once - baseline
  Demographics questionnaire (age, gender, education, disease duration)
Disease severity | Part III - once at baseline. Part I, II and IV - twice baseline and after 12 months
  Movement Disorders Society - Unified Parkinson's Disease Rating Scale part I-IV, with scores ranging from 0 to 272, in which the higher the score the worse symptoms are.
Disease status | Once - baseline
  Hoehn & Yahr stadia, ranging from 0-5, in which the higher the worse the disease status is.
Medication | Continuously over 12 months
  Medication intake diary
Balance - I | Once - baseline
  Mini-BESTest, ranging from 0 to 28, in which the higher the score the better the balance
Balance - II | Once - baseline
  Single leg stance test
Freezing of gait - I | Twice - baseline and after 12 months
  New freezing of gait questionnaire, ranging from 0 to 24, in which the higher the score the worse is the freezing of gait.
Freezing of gait - II | Once - baseline
  Rapid turns test
Cognition | Once - baseline
  Montreal Cognitive Assessment, with scores ranging from 0 to 30, in which the higher the better the cognition.
Sleep quality | Twice - baseline and after 12 months
  Pittsburgh Sleep Quality Index, with scores ranging from 0 to 21, in which the higher the worse the sleep quality.
Sleep quality and quantity | Once for a full week
  Sleep diary

CONTACTS AND LOCATIONS:
Overall Officials: Nienke M de Vries, Dr, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All data will be anonymized. The wearable sensor data will not be available for re-use and/or sharing.
Supporting Information: Analytic Code
Time Frame: After study completion.
Access Criteria: Access to the data will be granted for those performing research about Parkinson's disease.
URL: https://easy.dans.knaw.nl/ui/home